CLINICAL TRIAL: NCT02181192
Title: Postoperative Prostate Carcinoma Recurrence: Instant Radiotherapy Versus Radiotherapy With Additional Imaging With PSA Value >= 1
Brief Title: Point in Time of Radiotherapy for Patients With Biochemical Recurrent Prostate Carcinoma
Acronym: PROST-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROST-I
Record Dates: First submitted 2014-02-18; First posted 2014-07-03 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer; Recurrence
Keywords: biochemical recurrence; prostate carcinoma; prostate cancer; PSA; postoperative; radiotherapy; imaging diagnostic; PET/CT; social economic aspects; quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- delayed radiotherapy (Experimental): PET/CT and Radiotherapy after achievement of PSA marginal value Additive imaging
  Interventions: Device: PET/CT; Radiation: Radiotherapy after achievement of PSA marginal value
- instant radiotherapy (Active Comparator): Instant Radiotherapy according to guidelines
  Interventions: Radiation: Instant Radiotherapy according to guidelines

INTERVENTIONS:
Device: PET/CT — PET/CT
  Arms: delayed radiotherapy
Radiation: Instant Radiotherapy according to guidelines — Instant Radiotherapy according to guidelines
  Arms: instant radiotherapy
Radiation: Radiotherapy after achievement of PSA marginal value — Radiotherapy after achievement of PSA marginal value
  Arms: delayed radiotherapy

SUMMARY:
PSA-recurrence prostate carcinoma is associated with two general problems.

1. Localisation of PSA-recurrence is unconfident. In many cases it's not clear if a local, locoregional oder systemic relapse is available.
2. There is no standard therapy proved by randomised clinical trials. Recommended radiotherapy starting with PSA-value < 0.5 ng/ml according to german S3 guidelines is based on retrospective data.

These difficulties may lead to a therapy potentially not adapted to patients situation of disease.This study aims to randomised examine if an instant radiotherapy of prostate PSA-recurrence (PSA-value between 0.2 - 0.99 ng/ml) or a delayed radiotherapy with additional imaging (PSA value >= 1 ng/ml) including PET/CT and bone scintigraphy for reliable information about tumor location and expansion is beneficial regarding therapy efficiency, quality of life and social economic aspects.

ELIGIBILITY:
Inclusion Criteria:

* postoperative, biochemical recurrent prostate carcinoma with PSA value between 0.2 to 0.99 ng/ml
* prior irradiation
* comprehension of study protocol content and signed informed consent form
* minimum age 18 years

Exclusion Criteria:

* primary therapy of prostate carcinoma
* PSA value >= 1 ng/ml
* diagnosed distant metastases before randomisation (osseous or systemic)
* performed PET/CT before randomisation
* malignant slave tumor
* potent men that are not willing or are unable to apply consequent contraception
* ongoing drug- and/or alcohol abuse
* patients that are not willing or able to cooperate according to protocol
* patients in care
* patients that are not able to understand German language

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-07; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival according to PSA-value | at the end of follow-up period of 4 years
  Subjects in the control arm have an aftertreatment period of 5 years. Follow-up period of intervention arm ends after 3 to 5 years after radiotherapy. Duration depends on the surveillance period until marginal value is reached. This period is subtracted from maximum follow-up period of 5 years.

SECONDARY OUTCOMES:
frequency of PSA-persistence | at the end of therapy , an expected average of 6 weeks
frequency of changes in therapeutic strategies by additional diagnostics | at the end of therapy , an expected average of 6 weeks
analysis for radiation parameters, restricted to patients of initiating center | at the end of therapy , an expected average of 6 weeks
therapy and following costs for patients | time frame of 2 weeks before therapy starts; at the end of therapy , an expected average of 6 weeks; during follow-up each 3 months for the first 2 years, then each 6 months for the rest of follow-up period, an expected average of 2 further years
overall survival | at the end of therapy , an expected average of 6 weeks
quality of life and side effects | time frame of 2 weeks before therapy starts; at the end of therapy , an expected average of 6 weeks; during follow-up each 3 months for the first 2 years, then each 6 months for the rest of follow-up period, an expected average of 2 further years

CONTACTS AND LOCATIONS:
Overall Officials: Annedore Strnad, Dr. MHBA, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen; Rainer Fietkau, Dr., Study Director — Strahlenklinik, Universitätsklinikum Erlangen